CLINICAL TRIAL: NCT07141108
Title: Egenmonitorering Och Distansmonitorering av långvarig smärta i primärvården, användandet av Ett Digitalt Verktyg för Att ökad livskvalité
Brief Title: Self-monitoring and Remote Monitoring of Chronic Pain in Primary Care - Using a Digital Tool to Improve Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PD 2025-1
Record Dates: First submitted 2025-05-23; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Persistent Pain; Pain Management; Remote Monitoring
Keywords: chronic pain; pain management; persistent pain
MeSH Terms: conditions — Agnosia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital pain management Intervention Group (Experimental): Participants in this arm will use the Paindrainer® digital tool as part of their pain management strategy in primary care. Paindrainer® consists of a mobile app for self-monitoring of activity levels and symptoms, and a CARE portal for healthcare providers to support remote monitoring. The tool uses advanced neural networks to provide personalized feedback to help individuals plan and balance daily activities, aiming to enhance self-management and patient-provider communication. Standard care in primary care will continue in parallel. The study will evaluate the feasibility of implementing Paindrainer® in primary care settings and its potential to support long-term management of persistent pain conditions.
  Interventions: Device: Paindrainer Care system

INTERVENTIONS:
Device: Paindrainer Care system — Self management digital tool for chronic pain

SUMMARY:
Chronic pain impacts individuals, their families, and society significantly, yet specialist care resources are limited, with most patients managed in primary care. There is a need for tools that support self-management and improve resource allocation. This feasibility study evaluates the implementation of Paindrainer®, a CE-marked Class I digital tool, in primary care. Paindrainer® combines patient self-monitoring via an app with a healthcare provider portal (CARE) for remote monitoring. Using advanced neural networks, it offers personalized feedback to help patients plan and monitor daily activities and their impact on pain. The study aims to assess whether integrating this tool can enhance chronic pain management and patient quality of life.

DETAILED DESCRIPTION:
Long-term pain causes significant suffering to the individual, their loved ones and also entails high societal costs. In specialist care, constant development is underway through the implementation of new research and clinical findings. Patients' own efforts, decisions and strategies are a central and effective part of today's pain management. The importance of strengthening communication between patient and healthcare professionals is increasingly emphasised, as well as promoting the patient's ability to self-manage their situation.

More recently, behavior-modifying techniques have been integrated as complementary measures in the treatment of chronic pain. Despite this, a challenge remains for the healthcare system to create long-term sustainable outcomes for people with chronic pain.

The proportion of people with long-term pain who currently receive treatment in specialist care is very small, and the majority are treated in primary care instead. Resources for this patient group are insufficient and there is a great need for new tools for self- and remote monitoring that could improve the allocation of resources for this group.

This feasibility study aims to investigate whether a digital remote monitoring tool, Paindrainer®, can be implemented in primary care. The tool contains two parts, an app for the patient to use for their own monitoring of activity levels and symptoms, and the CARE portal, which is a remote monitoring tool for healthcare. The study will further explore how the implementation of this digital app in the existing treatment strategy can help address these challenges and improve care for people with chronic pain.

Paindrainer® is a CE marked class 1 product according to MDR and is based on advanced neural networks, which enables sophisticated calculations and takes into account more variables that affect the individual's pain experience and function than the human brain can handle. By using advanced calculations, Paindrainer provides continuous feedback to the patient, giving them a tool to plan and monitor their activities and understand how they affect each other.

This study will further investigate how Paindrainer® can support the individual to plan their activities in both "necessary" areas (such as daily chores, work, sleep) and other areas that are valuable to the individual (e.g. extracurricular activities, social and physical activities). By strengthening the patient's own role, Paindrainer is expected to increase the individual's quality of life and perceived health in both the short and long term.

ELIGIBILITY:
Inclusion Criteria:

Has pain that affects daily life and has lasted for more than 3 months

Is over 18 years old

Understands Swedish or English

Is motivated and willing to use a digital tool for self-monitoring of activity level and symptoms

Has no planned surgeries during the study period

Has knowledge of and access to using a smartphone or tablet

Exclusion Criteria:

Severe or acute mental illness, severe anxiety, or depression

Ongoing history of substance use disorder

Serious illness under active treatment

Pain related to malignancy

Currently involved in legal proceedings or ongoing litigation related to low back or neck pain

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of a Digital Self-Management Tool to Support Primary Care in Managing Persistent Pain | 12 weeks
  Through the use of logged daily activities the overall purpose of this study is to investigate how the digital tool Paindrainer® can support primary care in assisting individuals with persistent pain, reducing the impact of pain in daily life, and improving quality of life. The study focuses on evaluating the effectiveness and usability of Paindrainer® in supporting primary care efforts to provide adequate care, enhance continuity, and increase patient confidence in managing long-term pain conditions. The primary parameter to analyse is PROMSI Pain interference 6a and usability questioners

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life measured by the PROMIS-29 Profile | From baseline to 12 weeks
  The Patient-Reported Outcomes Measurement Information System 29-Item Profile (PROMIS-29) is a validated questionnaire designed to assess multiple domains of health-related quality of life. It includes 29 items covering seven key domains: Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, and Pain Interference, along with a single item for Pain Intensity. Each domain consists of four items rated on a 5-point Likert scale, except for Pain Intensity, which uses an 11-point numeric rating scale (0-10). Higher scores indicate more of the concept being measured (e.g., higher fatigue, higher social participation).
Change in Pain Acceptance | From baseline to 12 weeks
  The Chronic Pain Acceptance Questionnaire-9 (CPAQ-9) is a validated, shortened version of the original CPAQ, designed to measure an individual's acceptance of chronic pain. The CPAQ-9 assesses two key components: Activity Engagement (participation in life activities despite pain) and Pain Willingness (openness to experiencing pain without attempts to control or avoid it). The questionnaire consists of 9 items rated on a 7-point Likert scale, where higher scores indicate greater acceptance of chronic pain.
Change in Pain Catastrophizing measured by the Pain Catastrophizing Scale (PCS) | From baseline to 12 weeks
  The Pain Catastrophizing Scale (PCS) is a validated questionnaire used to assess catastrophic thinking related to pain, including elements of rumination, magnification, and feelings of helplessness. The scale consists of 13 items scored on a 5-point Likert scale. Higher scores indicate greater levels of pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Midlöv, Professor MD, Principal Investigator — Lunds Universitet
Locations (1):
- Lunds Universitet Centrum för Primärvårdsforskning (CPF) Institutionen för kliniska vetenskaper, Malmö, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (demographic information, primary and secondary outcomes) will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available starting 6 months after publication of primary results and will be accessible for 5 years thereafter.
Access Criteria: Qualified researchers with an approved proposal can request access via the study sponsor. Data will be shared through a secure data sharing platform.